CLINICAL TRIAL: NCT06265259
Title: Efficacy of the Use of Vasopressin as a Primary Vasoconstrictor in Critically Ill Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Vasiliki Tsolaki, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31-05-2023/25481
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Circulatory Shock
Keywords: noradrenaline; vasopressin; shock; multiorgan failure; SOFA score
MeSH Terms: conditions — Shock; Diabetes Insipidus; Multiple Organ Failure | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vasopresin Group (Experimental): Initiation of vasopressin as the first vasoactive agent (1 amp in 50 mlN/S) up to a maximum dose of 0.03 IU/min (2.3 ml/h). If the patient has MAP <65 mmHg then noradrenaline will be started.
  Interventions: Drug: Initiation of vasopressine as a first vasoconstrictive drug
- Noradrenaline group (Active Comparator): Initiation of noradrenaline first, up to 0,5 mcg/kg/min. If the patient has MAP <65 mmHg vasopressin will be started (maximum dose of 0.03 IU/min (2.3ml/h)]. If If the patient has MAP <65 mmHg, noradrenaline will be further escalated.
  Interventions: Drug: Initiation of noradrenaline as a first vasoconstrictive drug

INTERVENTIONS:
Drug: Initiation of vasopressine as a first vasoconstrictive drug — The group (arm 1) where vasopressin (1 amp in 50 mlN/S) (1st vasoconstrictor) will be administered first up to a maximum dose of 0.03 IU/min (2.3 ml/h) for the treatment of hemodynamic instability. Then, if the patient remains unstable, noradrenaline (2nd vasoconstrictor) will be started. The dose of vasopressin will not be increased further than the above mentioned limit.
  Other Names: Vasopressine, Empressin
  Arms: Vasopresin Group
Drug: Initiation of noradrenaline as a first vasoconstrictive drug — ii. In the group (arm 2) where the treatment of haemodynamic instability will be performed by first administering noradrenaline (1st vasoconstrictor) up to 0,5 mcg/kg/min and then, if the patient is still unstable, adding vasopressin (2nd vasoconstrictor) at a maximum dose of 0.03 IU/min (2.3ml/h). If haemodynamic instability persists, treatment will involve further increase of the noradrenaline dose.
  Other Names: Noradren, Levophed
  Arms: Noradrenaline group

SUMMARY:
Current guidelines recommend the inititaion of noradrenaline and if shock is refractory, then vasopressin should be administered. Data indicate that the earlier use of vasopressin may improve survival. Two large randomized controlled trial failed to prove a survival benefit from the early use of vasopressin. The present study will investigate the effect of an early initiation protocol of vasopressin (as the first vasoconstrictor drug) on the degree of multiorgan failure improvement and also on the course of sepsis (if in septic patients) versus early initiation of noradrenaline as first vasoconstrictor drug in hemodynamically unstable patients.

DETAILED DESCRIPTION:
1.2 Hypothesis - Literature Review The treatment of circulatory shock due to vasoparalysis in critically ill patients is based on the administration of fluids and vasopressors. In recent years a new vasopressor, vasopressin, has been recommended to be added to septic patients in need of low to moderate doses of noradrenaline to reduce the negative effects of circulating in elevated concentrations catecholamines. The aim of the present study is to investigate the degree of multiorganic failure improvement in patients with an early administration of vasopressin (as the first vasoconstrictor drug) versus noradrenaline on the outcome of critically ill patients in need of hemodynamic support with vasoactive drugs.

Vasopressin is an endogenous peptide that through V1 receptors causes selective vasoconstriction in non-vital organs and increases blood flow to the myocardium and brain. Vasopressin via V2 receptors causes vasodilation in coronary vessels as well as in cerebral vessels.

Noradrenaline (or norepinephrine) "is a potent peripheral vasoconstrictor which acts both on arterial and venous substrates (alpha-adrenergic effect) and as a cardiac inotropic stimulator. These effects result in an increase in systemic arterial pressure and blood flow in the coronary arteries".

Several studies have shown that the addition of vasopressin may allow the total norepinephrine / noradrenaline dose to be reduced. Vasopressin levels are thought to increase in the initial phase of shock in response to hypotension but then decrease over the following 48 to 72 hours resulting in relative vasopressin deficiency. However, a subgroup analysis in the Vasopressin and Septic Shock Trial (VASST) showed extremely low baseline vasopressin levels in patients with septic shock, so the lack of vasopressin is obvious. At the same time, the same subanalysis found a survival benefit in patients given vasopressin when the norepinephrine dose was less than 15 μg/min.

Two further studies showed that starting vasopressin very early (within four hours of initiating treatment with noradrenaline) in combination with noradrenaline: allowed earlier achievement and maintenance of Mean Arterial Pressure, improved organ function and led to a shorter length of hospital stay compared to noradrenaline. Rydz et al., showed that earlier initiation of vasopressin (within 7.3 h of starting noradrenaline) was associated with a greater likelihood of patients showing improvement in their multiorgan failure score and/or survival compared with those who had a delay in starting vasopressin.

The effect of administration of vasopressin as the first vasoconstrictor drug therefore seems to have not been assessed so far, whereas, in contrast, the literature estimates the effect of starting vasopressin in patients receiving low to moderate doses of noradrenaline. According to the existing data, it appears that vasopressin deficiency may occur as early as the early stages of septic shock. Also, the effect of vasopressin on patients with distribution shock other than septic patients, such as patients with a systemic inflammatory response as a consequence of brain injury (ischaemia, brain haemorrhage, head injury), has not been assessed.

For this reason, the present study will investigate the effect of an early initiation protocol of vasopressin (as the first vasoconstrictor drug) on the degree of multiorgan failure improvement and also on the course of sepsis (if in septic patients) versus early initiation of noradrenaline as first vasoconstrictor drug in hemodynamically unstable patients.

1.3 Research objectives of the study

Primary:

I. The primary endpoint of the study is to investigate the effect of early administration of vasopressin as the first vasoconstrictor drug followed by noradrenaline in hemodynamically unstable patients due to circulatory shock to the degree of multiorgan failure improvement as indicated by the Sequential Organ Failure Score (SOFA)) compared to patients in whom vasopressin is started after noradrenaline, according to existing guidelines. The degree of multiorgan failure will be assessed by recording the degree of multiorgan failure as assessed by the SOFA score. The recording will be done on days 0/ 3/ 5/ 7/ 10.

Secondary I. Duration of administration of vasoconstrictors, maximum daily dose. II. Assessment of the course of sepsis [recording of white blood cells, C-reactive protein (CRP), procalcitonin (PCT)]. Recording will be done on days 0/ 3/ 5/ 7/10.

III. Laboratory testing of urea - creatinine - transaminases - occlusive enzymes - total bilirubin - CPK-platelets and coagulation on days 0/ 7/ 14/ 28.

IV. Troponin and Brain Natriuretic Peptide B (BNP) values on days 0/ 3 / 5 / 7. V. Severity of renal impairment based on KDIGO 2022 criteria on the 3rd - 7th - 14th - 28th day of hospitalization.

VI. Fluid balance in the first 5 days. VIII. Need to use venovenous hemodialysis. IX. Days of mechanical ventilation. X. Number of septic episodes at 28 days. XI. Total length of stay in ICU XII. Mortality (28 days, ICU)

XIII. Recording of complications such as:

A) Ischaemic electrocardiographic changes. B) Arrhythmias (supraventricular tachycardia, atrial fibrillation, atrial flutter).

C) Incidence of paralytic ileus, episodes of ischaemic colitis (haemorrhagic stools, signs of ischaemic colitis and need for colonoscopy).

D) Ischaemia of limbs (how many fingers are ischaemic, where, to what extent). 1.4 Study design Randomised study. 1.5 Study population Patients who are hospitalized in the Intensive Care Unit, under mechanical ventilatory support and have circulatory failure and need to be administered vasoconstrictor drugs.

2. METHODS

1. Design - Study Protocol

The methodology to be followed will be a comparison between 2 cohorts of patients:

i. The group (arm 1) where vasopressin (1 amp in 50 mlN/S) (1st vasoconstrictor) will be administered first up to a maximum dose of 0.03 IU/min (2.3 ml/h) for the treatment of hemodynamic instability. Then, if the patient remains unstable, noradrenaline (2nd vasoconstrictor) will be started. The dose of vasopressin will not be increased further than the above mentioned limit.

ii. In the group (arm 2) where the treatment of haemodynamic instability will be performed by first administering noradrenaline (1st vasoconstrictor) up to 0,5 mcg/kg/min and then, if the patient is still unstable, adding vasopressin (2nd vasoconstrictor) at a maximum dose of 0.03 IU/min (2.3ml/h). If haemodynamic instability persists, treatment will involve further increase of the noradrenaline dose.

The goal is to achieve an average blood pressure of 65-75 mmHg. In each patient, the de-escalation will be applied first to the 2nd vasoconstrictor drug used in the arm to which it belongs and the 1st vasoconstrictor drug will be de-escalated last. In the event that a patient needs to be re-administered a vasoconstrictor (if he / she has been decompensated) then the first vasoconstrictor to be used will be the 1st vasoconstrictor administered in the arm to which he / she belongs.

2.1 Inclusion criteria All patients who have hemodynamic instability and distribution shock and require the administration of vasoconstrictor drugs after initial resuscitation. Patients include those with septic shock or systemic inflammatory reaction as a consequence of brain injury (ischaemia; brain haemorrhage, head injury).

2.2 Exclusion criteria

The patients excluded from this study are as follows:

* Patients under 18 years of age.
* Known heart failure (ejection fraction <35%)
* Recent acute myocardial infarction
* Pulmonary embolism 3. Ethical issues This clinical study will be conducted in accordance with the principles of the Declaration of Helsinki and will be carried out after approval by the Scientific Ethics Committee of the University General Hospital of Larissa.

With regard to the protection of patients' personal data, it is explicitly and categorically emphasized that their confidentiality and protection will be guaranteed. The study will be carried out respecting the anonymity of the participating patients, covering the full names with Arabic numbers (e.g. Patient 1, 2, etc.). The only people who will know which participant corresponds to which number will be the study investigators. Finally, the consent of the individual - or in case of the individual's incapacity - the consent of the next of kin, will be obtained for inclusion in the study.

4. DATA COLLECTION

During data collection, checks will be carried out on the following:

* Demographic characteristics (Age / Gender / Body Mass Index).
* Comorbidities. (Charlson Comorbidity Index - CCI)
* Cause of admission to the ICU.
* APACHE II (Acute Physiology and Chronic Health Evaluation II) Score
* SOFA (Sequential Organ Failure Assessment) Score during days 0 /3/ 5/ 7/ 10.
* Lactic acid course in the first 7 days (maximum value at 24 hours).
* Venous blood oxygen (SvO2) concentration changes in the first 7 days (maximum value at 24 hours).
* Average blood pressure (average value at 24 hours).
* Average daily urinary output.
* Renal function values on days (creatinine measurement) 0 / 3/ 5/ 7/ 10/ 14 / 28.
* Liver biochemistry values on days 0 / 3/ 5/ 7 / 10 / 14/ 28.
* Sodium on days 0/ 3/ 5/ 7/ 10/ 14/ 28.
* SOFA score on days 0/ 3/ 5/ 7/ 10.
* Albumin measurement 0/ 3/ 5 / 7/ 10.
* Cumulative dose/ maximum dose of vasopressin and noradrenaline on days of hospitalization and per day for the first 10 days of hospitalization.
* Days of vasoconstrictor administration and recording of the day of discontinuation of the second vasoconstrictor.
* Days off mechanical renal support during the 28-day period (CRRT-free days).
* Days off stage III, according to AKI, renal failure (d28).
* Adverse events (cardiovascular events, arrhythmias, limb ischemia, bowel ischemia).
* Mortality at 28 days.
* Mortality in the ICU. 5. EXPECTED RESULTS Improvement of multiorgan failure in patients with circulatory failure secondary to shock by using a vasoconstrictor drug administration protocol in which vasopressin is initiated as the first vasoconstrictor followed by noradrenaline, versus initiating noradrenaline as the primary vasoconstrictor.

ELIGIBILITY:
Inclusion Criteria:

• Shock (mean arterial pressure <65 mmHg) after initial resuscitation with fluids

Exclusion Criteria:

* Patients under 18 years of age.
* Known heart failure (ejection fraction <35%)
* Recent acute myocardial infarction
* Pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Multiorgan failure improvement assessment | 10 days
  Sequential Organ Failure Assessment score (min value 0, maximum value 24, with higher scores indicating worse patient status)

SECONDARY OUTCOMES:
Sepsis course | 10 days
  white blood cells
Sepsis course | 10 days
  C-reactive protein (CRP)
Sepsis course | 10 days
  procalcitonin (PCT)
Duration of administration of vasoconstrictors | 10 days
  Duration of administration of vasoconstrictors, maximum daily dose
laboratory tests | 28 days
  SGOT
laboratory tests | 28 days
  SGPT
laboratory tests | 28 days
  gGlutamile Transferase
laboratory tests | 28 days
  Alkaline Phoshatase
laboratory tests | 28 days
  Creatinophosphokinase
laboratory tests | 28 days
  total bilirubin
laboratory tests | 28 days
  urea
laboratory tests | 28 days
  creatinine
laboratory tests | 28 days
  Platelets
laboratory tests | 28 days
  Prothrombin time
laboratory tests | 28 days
  Partial thromboplastin time
Cardiac enzymes | 7 days
  Brain Natriuretic Peptide B (BNP)
Cardiac enzymes | 7 days
  Troponin
renal function | 28 days
  Severity of renal impairment based on KDIGO 2022 criteria
renal function | 5 days
  Fluid balance
renal function | 28 days
  Need for renal replacement therapy
Mechanical ventilation duration | 28 days
  IX. Days of mechanical ventilation
length of ICU stay | 90 DAYS
  Total days in ICU
28 day mortality | 28 days
  Mortality in 28 days
ICU mortality | 90 days
  ICU mortality
Adverse events | 28 days
  XIII. Recording of complications such as: A) Ischaemic electrocardiographic changes. B) Arrhythmias (supraventricular tachycardia, atrial fibrillation, atrial flutter). C) Incidence of paralytic ileus, episodes of ischaemic colitis (haemorrhagic stools, signs of ischaemic colitis and need for colonoscopy). D) Ischaemia of limbs (how many fingers are ischaemic, where, to what extent).

CONTACTS AND LOCATIONS:
Locations (1):
- General University Hospital of Larissa, Intensive Care Unit, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rydz AC, Elefritz JL, Conroy M, Disney KA, Miller CJ, Porter K, Doepker BA. EARLY INITIATION OF VASOPRESSIN REDUCES ORGAN FAILURE AND MORTALITY IN SEPTIC SHOCK. Shock. 2022 Oct 1;58(4):269-274. doi: 10.1097/SHK.0000000000001978. Epub 2022 Aug 16. PMID 36018257
- [Result] Hammond DA, Cullen J, Painter JT, McCain K, Clem OA, Brotherton AL, Chopra D, Meena N. Efficacy and Safety of the Early Addition of Vasopressin to Norepinephrine in Septic Shock. J Intensive Care Med. 2019 Nov-Dec;34(11-12):910-916. doi: 10.1177/0885066617725255. Epub 2017 Aug 18. PMID 28820036
- [Result] Sharshar T, Blanchard A, Paillard M, Raphael JC, Gajdos P, Annane D. Circulating vasopressin levels in septic shock. Crit Care Med. 2003 Jun;31(6):1752-8. doi: 10.1097/01.CCM.0000063046.82359.4A. PMID 12794416
- [Result] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Result] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Result] Hammond DA, Ficek OA, Painter JT, McCain K, Cullen J, Brotherton AL, Kakkera K, Chopra D, Meena N. Prospective Open-label Trial of Early Concomitant Vasopressin and Norepinephrine Therapy versus Initial Norepinephrine Monotherapy in Septic Shock. Pharmacotherapy. 2018 May;38(5):531-538. doi: 10.1002/phar.2105. Epub 2018 Apr 30. PMID 29600824